CLINICAL TRIAL: NCT02489630
Title: Low Dose Ketamine as an Adjunct to Opiates for Acute Pain in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08302015
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Acute Pain; Pain
MeSH Terms: conditions — Acute Pain; Pain | interventions — Ketamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): 0.1 mg/kg ketamine + opiate analgesic
  Interventions: Drug: Ketamine; Drug: opiate analgesic
- Placebo (Placebo Comparator): 0.1 mL/kg normal saline + opiate analgesic
  Interventions: Drug: Normal Saline; Drug: opiate analgesic

INTERVENTIONS:
Drug: Ketamine — 0.1mg/kg ketamine IV
  Other Names: Ketalar
  Arms: Ketamine
Drug: Normal Saline — 1ml/kg normal saline placebo
  Other Names: NS, saline
  Arms: Placebo
Drug: opiate analgesic — 0.1mg/kg dose of morphine (or morphine equivalent) at 30 min time intervals based on patient pain score or more frequently upon request

SUMMARY:
This study investigates the use of low doses of ketamine, along with opiate pain medication, is more effective at controlling the acute pain of patients in the emergency department than opiate pain medication alone. In addition, this study examines whether patients treated with low doses of ketamine, along with opiate pain medication, will require less opiate pain medication to control their pain, and whether these patients are equally happy with their pain control as patients who receive only opiate pain medication.

DETAILED DESCRIPTION:
This randomized, double blinded, placebo controlled study investigates the use of low-dose ketamine, in conjunction to standard opiate treatment, as compared to placebo plus standard opiate treatment, for acute painful conditions in the ED setting. The investigators hypothesize that patients treated with ketamine will require less opiate for similar levels of pain relief up to 2 hours from initiation of treatment, with similar levels of patient satisfaction and an acceptable side effect profile.

Once seen by a physician, potential patients will receive provider-determined opiate treatment for their painful condition, prior to the informed consent process to ensure that treatment is not delayed. Once identified for inclusion, patients will receive informed consent and, upon consent, will subsequently be randomized through block randomization into one of two study groups. Each study group will contain at least 50 subjects. Randomization will be determined using a table of random numbers, using a restricted randomization scheme to ensure roughly equal numbers in each group. Group assignments will be sealed in opaque envelopes to be opened sequentially by the investigators. Group assignments will not indicate whether it is the treatment or the control group. At this time (T0), an initial NRS-11 score will be obtained. The NRS-11 is an 11-point scale on which patients rate their level of pain from 0 ("no pain") to 10 ("worst pain imaginable"). If, after initial analgesic, pain level is <6, patients will be asked again in 15 min. If at this time it is still <6, they will not proceed in the study. The intervention group will receive 0.1 mg/kg of ketamine given over 1 minute, and the control group will receive an equivalent volume of normal saline; both groups will have received a provider-determined dose of opiate analgesia prior to enrollment. At thirty-minute intervals, subjects will be asked their level of pain, if they need more pain control and will be evaluated for the presence of side effects (hallucinations, dysphoria, weakness, diplopia, nausea, vomiting, dizziness, itching and bradypnea) as well as sedation as defined by Ramsay score of greater than 2. Repeat doses of pain medication will be given as 0.05 mg/kg morphine or equivalent dose of opioid analgesic. Total opiate dosage and number of repeat doses given at the end of 120 minutes will be recorded. At each time interval, as well as at the end of 120 minutes (T120), patient satisfaction with pain control will be recoded on the 4-point Likert scale, with 0 being "completely unsatisfied" and 3 being "very satisfied".

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years but less than 70 years old.
* Exhibiting pain defined on a numerical rating scale (NRS-11 [Farrar et al. 2001]) score of equal to or greater than 6 out of 10
* Deemed by the treating EM physician to require opioid analgesia.

Exclusion Criteria:

* Respiratory, hemodynamic or neurologic compromise, as determined by observation of signs of respiratory distress, systolic blood pressure less than 90 mmHg or systolic/diastolic blood pressure greater than 160/90, or a Glasgow -Coma Score less than 15.
* A history of chronic ventilation, dialysis or with previously diagnosed cirrhosis or hepatitis by istory.
* Active psychosis.
* Clinical intoxication.
* Known sensitivity to any study drug.
* An inability to understand the NRS-11 pain measurement scale.
* Presentation with headache or chest pain.
* Pregnancy.
* A lack of decision-making capacity.
* A pain score less than 6 on the NRS-11 scale.
* A concern by the treating physician or study personnel of current or prior history of narcotic abuse, or other secondary gain.
* Previously participated in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey R Heitz, MD, Principal Investigator — Physician

REFERENCES:
- [Background] Ahern TL, Herring AA, Stone MB, Frazee BW. Effective analgesia with low-dose ketamine and reduced dose hydromorphone in ED patients with severe pain. Am J Emerg Med. 2013 May;31(5):847-51. doi: 10.1016/j.ajem.2013.02.008. Epub 2013 Apr 18. PMID 23602757
- [Background] Beaudoin FL, Lin C, Guan W, Merchant RC. Low-dose ketamine improves pain relief in patients receiving intravenous opioids for acute pain in the emergency department: results of a randomized, double-blind, clinical trial. Acad Emerg Med. 2014 Nov;21(11):1193-202. doi: 10.1111/acem.12510. PMID 25377395
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Jennings PA, Cameron P, Bernard S, Walker T, Jolley D, Fitzgerald M, Masci K. Morphine and ketamine is superior to morphine alone for out-of-hospital trauma analgesia: a randomized controlled trial. Ann Emerg Med. 2012 Jun;59(6):497-503. doi: 10.1016/j.annemergmed.2011.11.012. Epub 2012 Jan 13. PMID 22243959
- [Background] Johansson P, Kongstad P, Johansson A. The effect of combined treatment with morphine sulphate and low-dose ketamine in a prehospital setting. Scand J Trauma Resusc Emerg Med. 2009 Nov 27;17:61. doi: 10.1186/1757-7241-17-61. PMID 19943920
- [Background] Kissin I, Bright CA, Bradley EL Jr. The effect of ketamine on opioid-induced acute tolerance: can it explain reduction of opioid consumption with ketamine-opioid analgesic combinations? Anesth Analg. 2000 Dec;91(6):1483-8. doi: 10.1097/00000539-200012000-00035. PMID 11094005

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 53 | 63
Completed | 51 | 61
Not Completed | 2 | 2
Not completed — Oversedation | 1 | 1
Not completed — Time to med. admin. > protocol limit | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 53 | 63 | 116
Age, Continuous [Mean (Full Range); unit: years] | 43.77 [18 to 69] | 41.43 [18 to 69] | 42.46 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 51
  Male | 31 | 34 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 51 | 63 | 114
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 63 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of Pain Control as Reported on the NRS-11
Description: Patient-reported pain scores on numerical rating scale (NRS) -11 pain scale (where 0 indicates no pain at all, 10 indicates the most severe pain). "Initial" group were patients enrolled and randomized in to the study, assessments were taken at the time of enrollment/randomization in to the study (up to 20 min prior to T=0). T = 0 min assessments were conducted at the time of medication administration (study allowed for an up to 20-minute delay in receiving study drug in order to retrieve study drug from secure storage, nursing documentation and patient verification prior to administration).
Time Frame: 20 min pre-medication administration, 0 min, 30 min, 60 min, 90 min, 120 min post medication administration
Population: Total number of study subjects; received intervention or placebo.
Measure: Mean (Standard Deviation); unit: Units on a scale (1-10)
Groups:
- Ketamine: Patients receiving study intervention
- Placebo: Patients not receiving study intervention
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 53 | 63
Units on a scale (1-10)
  Initial | 9.38 (0.97) | 9.44 (1.43)
  T = 0 min: number analyzed (Participants) | 52 | 62
  T = 0 min | 7.51 (1.53) | 8.10 (1.30)
  T = 30 min: number analyzed (Participants) | 50 | 61
  T = 30 min | 5.25 (2.58) | 2.27 (0.84)
  T = 60 min: number analyzed (Participants) | 45 | 54
  T = 60 min | 5.31 (2.79) | 6.18 (2.68)
  T = 90 min: number analyzed (Participants) | 38 | 48
  T = 90 min | 4.51 (2.63) | 6.21 (2.63)
  T = 120 min: number analyzed (Participants) | 25 | 28
  T = 120 min | 4.24 (2.95) | 5.68 (2.30)

2. Primary Outcome: Change in Patient Satisfaction With Pain Control on a 1-4 Likert Scale
Description: Patient-reported score regarding satisfaction with pain control, reported on a 4-point Likert scale (1-4, where 1 is the lowest satisfaction score possible and 4 is the highest satisfaction score possible). No data is reported for T = 0 min, as that assessment was conducted concurrently with initial medication dosing (since patients were at that point receiving their first pain control efforts, they could not yet assess their satisfaction with those efforts).
Time Frame: 0 min, 30 min, 60 min, 90 min, 120 min post medication administration
Population: Study subject-reported satisfaction with their pain control beginning at T = 30 minutes post-medication administration. Some study subjects were discharged, admitted or went to the operating room prior to this time point.
Measure: Mean (Standard Deviation); unit: Units on a scale (1-4)
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 50 | 61
Units on a scale (1-4)
  T = 30 min | 2.09 (0.88) | 2.27 (1.43)
  T = 60 min: number analyzed (Participants) | 45 | 55
  T = 60 min | 2.38 (0.76) | 2.33 (0.88)
  T = 90 min: number analyzed (Participants) | 38 | 48
  T = 90 min | 2.54 (0.65) | 2.38 (0.64)
  T = 120 min: number analyzed (Participants) | 25 | 28
  T = 120 min | 2.66 (0.67) | 2.52 (0.50)

3. Secondary Outcome: Difference in Opiate Dosage Between Study Arms in Morphine Equivalents
Description: Average difference in opiate dosage between study arms, calculated in morphine equivalents. "Initial" indicates at first dose of opioid administration, up to 20 mins prior to study drug administration, and from 0 min to 120 min after study drug administration.
Time Frame: 20 mins pre-medication administration, 0 min, 30 min, 60 min, 90 min, 120 min post medication administration
Population: Total number of patients receiving study intervention or placebo (less the two patients who were enrolled but did not receive medication within the protocol-defined time limit.
Measure: Mean (Standard Deviation); unit: Milligrams of Morphine Equivalent
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 52 | 62
Milligrams of Morphine Equivalent
  Initial Narcotic Dosage | 5.41 (2.77) | 5.83 (2.27)
  Total Narcotic Dosage | 9.95 (5.83) | 12.81 (6.81)

ADVERSE EVENTS:
Description: Collection approach for adverse events: regular investigator assessment.
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/63
Other Adverse Events (participants affected / at risk) | 0/53 | 0/63

LIMITATIONS AND CAVEATS:
This study was conducted in a busy ED in the general patient population, without special conditions, locations, or providers for study patients. The cohort includes subjects with chronic pain and long-term outpatient opioid use, as well as patients with new-onset acute pain; it is possible that the former patient population may react quite differently to the adjunctive ketamine usage than the latter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT02489630/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT02489630/SAP_001.pdf